CLINICAL TRIAL: NCT02858492
Title: A Multicenter, Randomized, Double-blind (Sponsor-unblinded), Placebo-controlled Study to Investigate the Safety and Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of GSK2982772 in Subjects With Moderate to Severe Rheumatoid Arthritis
Brief Title: Safety and Tolerability, Pharmacokinetics (PK), Pharmacodynamics (PD) and Efficacy of Repeat Doses of GSK2982772 in Subjects With Moderate to Severe Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 203168; 2016-000912-13 (EudraCT Number)
Record Dates: First submitted 2016-07-20; First posted 2016-08-08 (Estimated); Results first posted 2019-11-01 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Arthritis, Rheumatoid
Keywords: efficacy; safety; pharmacokinetics; pharmacodynamics; Rheumatoid Arthritis; autoimmune
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GSK2982772

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects receiving GSK2982772 60 mg (Experimental): Enrolled subjects will receive GSK2982772 60 mg thrice daily (approximately 8 hours apart) for 84 days.
  Interventions: Drug: GSK2982772 60 mg
- Subjects receiving Placebo (Experimental): Enrolled subjects will receive placebo thrice daily (approximately 8 hours apart) for 84 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2982772 60 mg — GSK2982772 is available as a 30 mg white to almost white, round film coated tablet which will be administered as two tablets thrice daily as directed.
  Arms: Subjects receiving GSK2982772 60 mg
Drug: Placebo — Placebo is available as a white to almost white, round film coated tablet which will be administered as two tablets thrice daily as directed.
  Arms: Subjects receiving Placebo

SUMMARY:
This study is the first study with GSK2982772, a receptor-interacting protein-1 (RIP1) kinase inhibitor, in subjects with moderate to severe RA who are currently being treated with disease modifying anti-rheumatic drugs (DMARDs). The primary objective of the study is to investigate the safety and tolerability of repeat oral doses of GSK2982772 in subjects with moderate to severe RA. In addition to the PK, a number of experimental and clinical endpoints will be employed to obtain information on the PD, and preliminary efficacy in subjects with active RA. Although no formal hypothesis will be tested, these endpoints will enable a broader understanding of the mechanism of action and potential for clinical efficacy of GSK2982772 in RA. After a screening period of up to 30 days, approximately 24 subjects will be randomized to receive either GSK2982772 or placebo for 84 days (12 weeks), followed by a follow-up period (28 days). The total duration of participation in the study will be approximately 20 weeks from screening to the last study visit.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 75 years of age inclusive, at the time of signing the informed consent.
* Subjects that do not have any medical conditions, other than moderate to severe RA, that in the opinion of the Investigator put the subject at unacceptable risk or interfere with study assessments or integrity of the data. These medical conditions should be stable at the time of screening and are expected to remain stable for the duration of the study.
* Subject has had a confirmed diagnosis of rheumatoid arthritis according to the revised 2010 ACR-EULAR classification criteria.
* Disease duration of >=12 weeks (time from onset of patient-reported symptoms of either pain or stiffness or swelling in hands, feet or wrists) at screening.
* Swollen joint count of >=4 (28-joint count) and tender joint count >=4 (28-joint count) at screening.
* Subject has a DAS28 CRP disease activity score of >= 3.2 and CRP >= 5.0 mg/liter (L) (>=4.76 nanomole (nmol)/L) at screening.
* Subject must have received at least 12 weeks of non-biologic DMARD monotherapy or MTX/DMARD combination therapy prior to screening and must be on stable dose throughout the study.
* Subject is naive to any biological therapies for RA or subject may have had previous exposure to a single anti-tumor necrosis factor (TNF) biologic agent which was discontinued for reasons other than primary non-response more than 8 weeks (or 5 half lives whichever is longer) from first dose.
* For subjects who have consented to synovial joint biopsy:

  • Subject has an involved knee, wrist, or ankle suitable for biopsy, as assessed by a rheumatologist at screening.
* A body mass index (BMI) within range of 18.5 - 35 kilogram/meter^2 (Kg/m^2) (inclusive) at screening.
* Male and female subjects Males: Male subjects with female partners of child bearing potential must comply with the contraception requirements specified in the protocol.

Females: A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotropin [HCG] test), not lactating, and at least one of the following conditions applies:

* Non-reproductive potential as defined as pre-menopausal females with either documented tubal ligation or Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion or Hysterectomy or Documented Bilateral Oophorectomy. For Postmenopausal females as 12 months of spontaneous amenorrhea in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment..
* Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication and until at least 30 days after the last dose of study medication and completion of the follow-up visit.

  * The Investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
  * Capable of giving signed informed consent as described in the protocol which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* Subject with a positive anti-double stranded deoxyribonucleic acid (DNA [anti-dsDNA]) and confirmed diagnosis of systemic lupus erythematosus (SLE).
* Subject with current history of Suicidal Ideation Behavior (SIB) as measured using the Columbia Suicide Severity Rating Scale (C-SSRS) or a history of attempted suicide.
* An active infection, or a history of infections as follows:

  * Hospitalization for treatment of infection within 60 days before first dose (Day 1).
  * Currently on any suppressive therapy for a chronic infection (such as pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria).
  * Use of parenteral (intravenous [IV] or intramuscular) antibiotics (antibacterials, antivirals, antifungals, or antiparasitic agents) for an infection within 60 days before first dose.
  * A history of opportunistic infections within 1 year of screening (e.g. pneumocystis jirovecii, cytomegalovirus [CMV] pneumonitis, aspergillosis). This does not include infections that may occur in immunocompetent individuals, such as fungal nail infections or vaginal candidiasis, unless it is of an unusual severity or recurrent nature.
  * Recurrent or chronic infection or other active infection that, in the opinion of the Investigator might cause this study to be detrimental to the patient.
  * History of Tuberculosis (TB), irrespective of treatment status.
  * A positive diagnostic TB test at screening defined as a positive QuantiFERON-TB Gold test or T-spot test. In cases where the QuantiFERON or T-spot test is indeterminate, the subject may have the test repeated once, but they will not be eligible for the study unless the second test is negative. In cases where the QuantiFERON or T-spot test is positive, but a locally-read follow up chest x-ray, shows no evidence of current or previous pulmonary tuberculosis, the subject may be eligible for the study at the discretion of the Investigator and GSK Medical Monitor.
* Electrocardiogram QT interval corrected for heart rate (QTc) > 450 milliseconds (msec) or QTc > 480 msec for subjects with bundle branch block at screening.

The QTc is the QT interval corrected for heart rate according to either Bazett's formula (QTcB), Fridericia's formula (QTcF), or another method, machine or manual over read. The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined and documented prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QTc for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trial. For purposes of data analysis, QTcB, QTcF, another QT correction formula, or a composite of available values of QTc will be used.

* Alanine aminotransferase (ALT) >2x upper limit of normal (ULN) and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent) at screening.
* Current active or chronic history of liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Current or history of renal disease or estimated glomerular filtration rate (GFR) by Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI) calculation <60 milliliter (mL)/minute (min)/1.73 m^2 at screening.
* Hereditary or acquired immunodeficiency disorder, including immunoglobulin deficiency.
* A major organ transplant (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/marrow transplant.
* Any planned surgical procedures including surgical joint procedures (e.g., intra-articular, tendon sheath, or bursal corticosteroid injections) during the study.
* A history of malignant neoplasm within the last 5 years, except for adequately treated non-metastatic cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix that has been fully treated and shows no evidence of recurrence.
* Has undergone surgery including synovectomy or arthroplasty on the joint chosen for biopsy and/or magnetic resonance imaging (MRI).
* The subject has a history of any other joint disease other than RA at the knee, wrist or ankle joint chosen for biopsy and/or MRI (e.g., gout, pseudogout, osteoarthritis).
* Has undergone intra-articular corticosteroid injection, arthrocentesis or synovial biopsy on any joint within 6 weeks of screening.
* A known allergy to lidocaine or other local anesthetics (only applies to subjects who consent for synovial biopsy procedures).
* Contraindication to MRI scanning (as assessed by local MRI safety questionnaire) which includes but are not limited to:

  * Intracranial aneurysm clips (except SugitaTM) or other metallic objects,
  * History of intra-orbital metal fragments that have not been removed by a medical professional.
  * Pacemakers or other implanted cardiac rhythm management devices and non-MR compatible heart valves,
  * Inner ear implants,
  * History of claustrophobia which may impact participation.
* The subject has received treatment with the prohibited therapies listed in the protocol, or changes to those treatments, within the prescribed timeframe.

  • Other medications (including vitamins, herbal and dietary supplements) will be considered on a case-by-case basis, and will be allowed if in the opinion of the Investigator the medication will not interfere with the study procedures or compromise subject safety.
* History of alcohol or drug abuse that would interfere with the ability to comply with the study.
* History of sensitivity to any of the study treatments, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation.
* Received a live or attenuated vaccine within 30 days of randomization or plan to receive a vaccination during the study until half-lives (or 2 days) plus 30 days after receiving GSK2982772.
* Contraindication to gadolinium contrast agent in accordance with local guidelines.
* The subject has participated in a clinical trial and has received an investigational product within 30 days or 5 half-lives, whichever is longer before the first dose of study medication, or plans to take part in another clinical trial at the same time as participating in this clinical trial.
* Hemoglobin <9 grams/deciliter (g/dL);hematocrit <30 percent, white blood cell count =<3,000/millimeter^3 (mm^3) (=<3.0 x 10^9/L); platelet count =<100,000/ microliter (μL) (=<100 x 10^9/L); absolute neutrophil count =<1.5 x 10^9/L at screening. For subjects recruited in Germany: hemoglobin <11 g/dL at screening.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. As potential for and magnitude of immunosuppression with this compound is unknown, subjects with presence of hepatitis B core antibody (HBcAb) should be excluded.
* A positive serology for human immunodeficiency virus (HIV) 1 or 2 at screening.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 3 months.
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first dose.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- Germany (2):
  - GSK Investigational Site, Rendsburg, Schleswig-Holstein
  - GSK Investigational Site, Berlin
- Italy (2):
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Verona, Veneto
- Poland (5):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Świdnik
  - GSK Investigational Site, Warsaw
- Russia (2):
  - GSK Investigational Site, Ulyanovsk
  - GSK Investigational Site, Yaroslavl
- Spain (3):
  - GSK Investigational Site, Málaga, Andalusia
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Barcelona
- United Kingdom (2):
  - GSK Investigational Site, Southampton, Hampshire
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20827

REFERENCES:
- [Background] Weisel K, Berger S, Thorn K, Taylor PC, Peterfy C, Siddall H, Tompson D, Wang S, Quattrocchi E, Burriss SW, Walter J, Tak PP. A randomized, placebo-controlled experimental medicine study of RIPK1 inhibitor GSK2982772 in patients with moderate to severe rheumatoid arthritis. Arthritis Res Ther. 2021 Mar 16;23(1):85. doi: 10.1186/s13075-021-02468-0. PMID 33726834

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study evaluated safety, pharmacokinetics (PK), pharmacodynamics (PD), and efficacy of GSK2982772 in participants with rheumatoid arthritis (RA). Participants were randomly assigned to receive either GSK2982772 60 milligram (mg) or placebo to be taken orally twice daily (BID) or three times daily (TID) for 84 days.
Pre-assignment Details: A total of 99 participants were screened, of them, 47 participants were screen failures and 52 participants were enrolled. Of them, 51 participants received study treatment. One participant was enrolled in the study but never received study treatment as eligibility criteria for dose was not met.
Groups:
- Placebo BID: Participants received placebo orally twice daily (BID) for 84 days (12 weeks). Participants received methotrexate for the treatment of RA during conduct of the study, if required.
- Placebo TID: Participants received placebo orally three times daily (TID) (approximately 8 hours apart) for 84 days (12 weeks). Participants received methotrexate for the treatment of RA during conduct of the study, if required.
- GSK2982772 60 mg BID: Participants received GSK2982772 orally twice daily (BID) for 84 days (12 weeks). Participants received methotrexate for the treatment of RA during conduct of the study, if required.
- GSK2982772 60 mg TID: Participants received GSK2982772 orally three times daily (TID) (approximately 8 hours apart) for 84 days (12 weeks). Participants received methotrexate for the treatment of RA during conduct of the study, if required.
Period: Overall Study
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Started | 3 | 15 | 5 | 28
Completed | 3 | 14 | 5 | 22
Not Completed | 0 | 1 | 0 | 6
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 3
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Protocol defined stopping criteria | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID | Total
Number analyzed (Participants) | 3 | 15 | 5 | 28 | 51
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.3 (4.93) | 53.1 (7.80) | 53.6 (7.86) | 55.0 (11.25) | 54.2 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 13 | 4 | 23 | 42
  Male | 1 | 2 | 1 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0 | 0 | 0 | 1 | 1
  White-White/Caucasian/European Heritage | 3 | 15 | 5 | 27 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-serious Adverse Events (nSAEs) and Serious Adverse Events (SAEs) as a Measure of Safety and Tolerability
Description: An AE was any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly or birth defect or any other situation according to medical or scientific judgment was categorized as SAE. Number of participants with any nSAE or SAE are presented.
Time Frame: Up to Day 112
Population: Safety Population comprised of all participants who received at least one dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 15 | 5 | 28
Participants
  Any nSAEs | 3 | 10 | 3 | 16
  Any SAEs | 0 | 0 | 0 | 2

2. Primary Outcome: Number of Participants With Worst Case Clinical Chemistry Parameters of Potential Clinical Importance (PCI)
Description: Clinical chemistry parameters included alanine amino transferase (ALT), albumin, alkaline phosphatase, aspartate amino transferase (AST), calcium, creatinine, glucose, potassium, sodium and total bilirubin. PCI ranges were ALT(high): >=2*Upper limit of Normal(ULN) units per liter(U/L), albumin(low): 30 millimoles per liter(mmol/L), alkaline phosphatase(high): >=2*ULN U/L, AST(high): >=2*ULN U/L, calcium: <2(low) or >2.75 mmol/L(high), creatinine (high): increase from Baseline >44.25 mmol/L, glucose: <3(low) or >9 mmol/L(high), potassium: <3(low) or >5.5 mmol/L(high), sodium: <130(low) or >150 mmol/L(high) and total bilirubin(high): >=1.5*ULN micromoles per liter(µmol/L). Participants were counted in the worst case category if their value changes (to low or to high), unless there is no change in their category. Only those clinical chemistry parameters with PCI values (to low and to high) have been presented.
Time Frame: Up to Day 112
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 15 | 5 | 28
Participants
  ALT; To low | 0 | 0 | 0 | 0
  ALT; To high | 0 | 0 | 0 | 2
  Albumin; To low | 0 | 0 | 0 | 0
  Albumin; To high | 0 | 0 | 0 | 0
  Alkaline phosphatase; To Low | 0 | 0 | 0 | 0
  Alkaline phosphatase; To high | 0 | 0 | 0 | 0
  AST; To low | 0 | 0 | 0 | 0
  AST; To high | 0 | 0 | 0 | 1
  Calcium; To low | 0 | 0 | 0 | 0
  Calcium; To high | 0 | 0 | 0 | 0
  Creatinine; To low | 0 | 0 | 0 | 0
  Creatinine; To high | 0 | 0 | 0 | 0
  Glucose; To low | 0 | 1 | 0 | 0
  Glucose; To high | 0 | 1 | 0 | 1
  Potassium; To low | 0 | 0 | 0 | 0
  Potassium; To high | 0 | 0 | 0 | 1
  Sodium; To low | 0 | 0 | 0 | 0
  Sodium; To high | 0 | 0 | 0 | 0
  Total bilirubin; To low | 0 | 0 | 0 | 0
  Total bilirubin; To high | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Worst Case Hematology Parameters of PCI
Description: Hematology parameters included hematocrit, hemoglobin, lymphocytes, platelet counts, total neutrophils and white blood cells (WBCs). PCI ranges were < 0.075 (decrease from baseline) or >0.54 proportion of red blood cells in blood (high) for hematocrit, <25 (low) or >180 grams per liter (g/L) (high) for hemoglobin, <0.8 x10^9 cells per liter (cells/L) for lymphocytes (low), <100 (low) or >550 x10^9 cells/L(high) for platelets, <1.5 x10^9 cells/L (low) for total neutrophils and < 3 (low) or >20 x10^9 cells/L (high) for WBCs. Participants were counted in the worst case category that their value changes (to low or to high), unless there is no change in their category. Only those hematology parameters with PCI values (to low and to high) have been presented.
Time Frame: Up to Day 112
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 15 | 5 | 28
Participants
  Hematocrit; To low | 0 | 0 | 0 | 0
  Hematocrit; To high | 0 | 0 | 0 | 0
  Hemoglobin; To low | 0 | 0 | 0 | 0
  Hemoglobin; To high | 0 | 0 | 0 | 0
  Lymphocytes; To Low | 2 | 1 | 0 | 1
  Lymphocytes; To high | 0 | 0 | 0 | 0
  Platelet count; To low | 0 | 0 | 0 | 0
  Platelet count; To high | 0 | 0 | 0 | 0
  Total neutrophils; To low | 0 | 0 | 0 | 1
  Total neutrophils; To high | 0 | 0 | 0 | 0
  WBC; To low | 0 | 0 | 0 | 1
  WBC; To high | 0 | 1 | 0 | 0

4. Primary Outcome: Number of Participants With Worst Case Any Increase in Urinalysis Results Post-Baseline Relative to Baseline by Dipstick Method
Description: Urine samples were collected to assess glucose, ketones, occult blood and protein by dipstick method. The dipstick test gave results in a semi-quantitative manner, and results for urinalysis parameters glucose, ketones, occult blood and protein were categorized as 'any increase from Baseline', which imply any increase in their concentrations in the urine sample. Only participants with worst case any increase from Baseline values are presented.
Time Frame: Up to Day 112
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 15 | 5 | 28
Participants
  Glucose; Any increase | 0 | 0 | 0 | 0
  Ketones; Any increase | 1 | 3 | 3 | 6
  Occult blood; Any increase | 0 | 6 | 1 | 8
  Protein; Any increase | 1 | 2 | 0 | 6

5. Primary Outcome: Number of Participants With Worst Case Any Increase in Urinalysis Results Post-Baseline Relative to Baseline by Microscopy Method
Description: Urine samples were collected to assess glucose, ketones, occult blood and protein by dipstick method. Microscopy was performed only on urine samples showing an abnormality on the dipstick. Microscopy was performed for hyaline casts, red blood cells and white blood cells. Results for microscopy parameters hyaline casts, red blood cells and white blood cells were categorized as 'any increase from Baseline', which imply any increase in their count in the urine sample. Only participants with worst case any increase from Baseline values are presented.
Time Frame: Up to Day 112
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 2 | 7 | 1 | 11
Participants
  Hyaline casts;any increase;n=0,1,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Hyaline casts;any increase;n=0,1,0,0 |  | 1 |  |
  Red blood cells;any increase;n=2,7,1,11 | 1 | 5 | 1 | 8
  White blood cells;any increase;n=2,7,1,11 | 2 | 5 | 1 | 7

6. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Heart Rate at Indicated Time Points
Description: 12- lead ECG was measured on each day using an ECG machine that automatically calculated the heart rate and measured PR interval, QRS duration, QT interval, QT interval corrected for heart rate according to either Bazett's formula (QTcB) and QT interval corrected for heart rate according to Fridericia's formula (QTcF). ECG was measured in semi-supine or supine position after 5 minutes rest. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline (Day 1 pre-dose), Days 8, 15, 29, 43, 57, 71 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 14 | 5 | 24
Beats per minute
  Day 8; n=3,14,5,23: number analyzed (Participants) | 3 | 14 | 5 | 23
  Day 8; n=3,14,5,23 | 7.0 (5.57) | 1.1 (10.68) | 0.6 (7.09) | 0.6 (7.55)
  Day 15; n=3,14,5,24 | 0.7 (2.08) | -0.3 (11.64) | -4.6 (4.16) | 1.0 (9.94)
  Day 29; n=3,14,5,22: number analyzed (Participants) | 3 | 14 | 5 | 22
  Day 29; n=3,14,5,22 | 2.7 (4.93) | -1.4 (8.27) | -5.8 (13.66) | 1.3 (9.14)
  Day 43; n=3,13,5,23: number analyzed (Participants) | 3 | 13 | 5 | 23
  Day 43; n=3,13,5,23 | -0.7 (7.57) | -3.5 (9.73) | -6.0 (7.35) | -0.2 (10.86)
  Day 57; n=3,13,5,22: number analyzed (Participants) | 3 | 13 | 5 | 22
  Day 57; n=3,13,5,22 | -3.7 (10.69) | -2.4 (8.79) | -4.2 (8.58) | 0.7 (9.75)
  Day 71; n=3,13,5,22: number analyzed (Participants) | 3 | 13 | 5 | 22
  Day 71; n=3,13,5,22 | 0.3 (9.29) | -3.0 (12.08) | -7.6 (7.73) | 0.3 (9.32)
  Day 85; n=3,13,5,21: number analyzed (Participants) | 3 | 13 | 5 | 21
  Day 85; n=3,13,5,21 | -1.7 (5.69) | -4.1 (11.51) | -2.4 (4.72) | -1.4 (9.12)

7. Primary Outcome: Change From Baseline in ECG PR Interval, QRS Duration, QT Interval, QTcB and QTcF at Indicated Time Points
Description: 12- lead ECG was measured on each day using an ECG machine that automatically calculated the heart rate and measured PR interval, QRS duration, QT interval QTcB and QTcF. ECG was measured in semi-supine or supine position after 5 minutes rest. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline (Day 1 pre-dose), Days 8, 15, 29, 43, 57, 71 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Millisecond
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 14 | 5 | 24
Millisecond
  PR interval; Day 8; n=3,14,5,23: number analyzed (Participants) | 3 | 14 | 5 | 23
  PR interval; Day 8; n=3,14,5,23 | -0.3 (14.36) | -1.9 (26.35) | -6.4 (19.98) | 0.8 (18.84)
  PR interval; Day 15; n=3,14,5,24 | 6.3 (12.66) | 0.6 (29.94) | -2.0 (23.10) | 3.0 (15.71)
  PR interval; Day 29; n=3,14,5,22: number analyzed (Participants) | 3 | 14 | 5 | 22
  PR interval; Day 29; n=3,14,5,22 | 5.3 (24.01) | -3.5 (32.15) | -0.2 (22.66) | -6.9 (28.00)
  PR interval; Day 43; n=3,13,5,23: number analyzed (Participants) | 3 | 13 | 5 | 23
  PR interval; Day 43; n=3,13,5,23 | 2.0 (17.35) | 6.5 (14.44) | 2.4 (5.41) | 6.6 (15.69)
  PR interval; Day 57; n=3,13,5,22: number analyzed (Participants) | 3 | 13 | 5 | 22
  PR interval; Day 57; n=3,13,5,22 | -12.0 (5.29) | 5.8 (21.75) | 5.0 (6.36) | 4.1 (17.51)
  PR interval; Day 71; n=3,13,5,22: number analyzed (Participants) | 3 | 13 | 5 | 22
  PR interval; Day 71; n=3,13,5,22 | 1.0 (17.78) | 1.2 (18.65) | 2.2 (23.92) | 0.8 (15.06)
  PR interval; Day 85; n=3,13,5,21: number analyzed (Participants) | 3 | 13 | 5 | 21
  PR interval; Day 85; n=3,13,5,21 | 1.3 (10.02) | 6.2 (15.38) | -0.2 (5.26) | 0.4 (10.29)
  QRS duration; Day 8; n=3,14,5,23: number analyzed (Participants) | 3 | 14 | 5 | 23
  QRS duration; Day 8; n=3,14,5,23 | -4.7 (5.03) | -3.3 (10.75) | 8.2 (10.33) | 3.7 (12.97)
  QRS duration; Day 15; n=3,14,5,24 | -3.3 (4.16) | -3.1 (10.50) | -1.2 (7.26) | 1.1 (6.89)
  QRS duration; Day 29; n=3,14,5,22: number analyzed (Participants) | 3 | 14 | 5 | 22
  QRS duration; Day 29; n=3,14,5,22 | -1.3 (3.79) | -2.1 (10.89) | 0.4 (5.03) | -0.5 (9.01)
  QRS duration; Day 43; n=3,13,5,23: number analyzed (Participants) | 3 | 13 | 5 | 23
  QRS duration; Day 43; n=3,13,5,23 | -3.3 (5.51) | -1.1 (9.90) | 3.6 (8.29) | 0.3 (10.48)
  QRS duration; Day 57; n=3,13,5,22: number analyzed (Participants) | 3 | 13 | 5 | 22
  QRS duration; Day 57; n=3,13,5,22 | -6.0 (6.00) | -4.0 (5.90) | 3.2 (9.34) | 1.0 (18.33)
  QRS duration; Day 71; n=3,13,5,22: number analyzed (Participants) | 3 | 13 | 5 | 22
  QRS duration; Day 71; n=3,13,5,22 | -10.0 (7.55) | -0.2 (6.68) | 4.6 (12.26) | -0.5 (8.31)
  QRS duration; Day 85; n=3,13,5,21: number analyzed (Participants) | 3 | 13 | 5 | 21
  QRS duration; Day 85; n=3,13,5,21 | -7.3 (11.37) | -1.0 (9.07) | 3.4 (8.68) | 1.5 (10.68)
  QT interval; Day 8; n=3,14,5,23: number analyzed (Participants) | 3 | 14 | 5 | 23
  QT interval; Day 8; n=3,14,5,23 | -25.7 (6.11) | 6.4 (40.17) | -14.2 (22.49) | -1.0 (35.97)
  QT interval; Day 15; n=3,14,5,24 | 2.7 (11.02) | 20.7 (34.85) | 0.0 (21.12) | -4.5 (25.27)
  QT interval; Day 29; n=3,14,5,22: number analyzed (Participants) | 3 | 14 | 5 | 22
  QT interval; Day 29; n=3,14,5,22 | -9.3 (17.67) | 7.6 (25.03) | -5.6 (22.37) | 5.5 (31.49)
  QT interval; Day 43; n=3,13,5,23: number analyzed (Participants) | 3 | 13 | 5 | 23
  QT interval; Day 43; n=3,13,5,23 | -12.7 (28.10) | 18.5 (38.73) | 1.0 (20.74) | 0.6 (29.36)
  QT interval; Day 57; n=3,13,5,22: number analyzed (Participants) | 3 | 13 | 5 | 22
  QT interval; Day 57; n=3,13,5,22 | 12.3 (30.04) | 13.6 (41.48) | 2.4 (22.78) | -1.8 (36.44)
  QT interval; Day 71; n=3,13,5,22: number analyzed (Participants) | 3 | 13 | 5 | 22
  QT interval; Day 71; n=3,13,5,22 | -9.3 (33.98) | 13.8 (32.50) | 10.2 (28.71) | -2.1 (22.06)
  QT interval; Day 85; n=3,13,5,21: number analyzed (Participants) | 3 | 13 | 5 | 21
  QT interval; Day 85; n=3,13,5,21 | -0.3 (14.50) | 17.2 (32.16) | -3.2 (14.60) | 3.0 (17.28)
  QTcB; Day 8; n=2,14,5,22: number analyzed (Participants) | 2 | 14 | 5 | 22
  QTcB; Day 8; n=2,14,5,22 | -12.1 (8.34) | 10.5 (46.28) | -10.3 (14.09) | 0.7 (33.20)
  QTcB; Day 15; n=2,14,5,23: number analyzed (Participants) | 2 | 14 | 5 | 23
  QTcB; Day 15; n=2,14,5,23 | 7.2 (7.18) | 22.9 (46.10) | -12.9 (17.59) | -0.9 (19.63)
  QTcB; Day 29; n=2,14,5,21: number analyzed (Participants) | 2 | 14 | 5 | 21
  QTcB; Day 29; n=2,14,5,21 | -2.4 (7.96) | 4.4 (25.73) | -21.2 (29.58) | 10.3 (29.02)
  QTcB; Day 43; n=2,13,5,22: number analyzed (Participants) | 2 | 13 | 5 | 22
  QTcB; Day 43; n=2,13,5,22 | -13.0 (14.51) | 9.1 (37.18) | -14.2 (14.64) | 0.6 (27.77)
  QTcB; Day 57; n=2,13,5,21: number analyzed (Participants) | 2 | 13 | 5 | 21
  QTcB; Day 57; n=2,13,5,21 | -1.5 (1.83) | 7.5 (38.73) | -7.0 (11.67) | 1.1 (47.85)
  QTcB; Day 71; n=2,13,5,21: number analyzed (Participants) | 2 | 13 | 5 | 21
  QTcB; Day 71; n=2,13,5,21 | -9.3 (16.59) | 4.6 (34.77) | -11.0 (16.47) | -1.1 (20.55)
  QTcB; Day 85; n=2,13,5,20: number analyzed (Participants) | 2 | 13 | 5 | 20
  QTcB; Day 85; n=2,13,5,20 | 4.2 (15.78) | 7.0 (32.09) | -9.1 (12.42) | -0.7 (17.51)
  QTcF; Day 8; n=2,14,5,22: number analyzed (Participants) | 2 | 14 | 5 | 22
  QTcF; Day 8; n=2,14,5,22 | -16.0 (3.35) | 9.0 (42.58) | -11.4 (14.05) | 0.3 (33.04)
  QTcF; Day 15; n=2,14,5,23: number analyzed (Participants) | 2 | 14 | 5 | 23
  QTcF; Day 15; n=2,14,5,23 | 7.5 (7.65) | 22.2 (39.68) | -8.4 (18.00) | -2.3 (17.61)
  QTcF; Day 29; n=2,14,5,21: number analyzed (Participants) | 2 | 14 | 5 | 21
  QTcF; Day 29; n=2,14,5,21 | -3.3 (13.16) | 5.6 (22.87) | -15.6 (18.24) | 8.7 (27.77)
  QTcF; Day 43; n=2,13,5,22: number analyzed (Participants) | 2 | 13 | 5 | 22
  QTcF; Day 43; n=2,13,5,22 | -13.5 (23.40) | 12.4 (35.37) | -8.7 (13.81) | 0.7 (25.16)
  QTcF; Day 57; n=2,13,5,21: number analyzed (Participants) | 2 | 13 | 5 | 21
  QTcF; Day 57; n=2,13,5,21 | 5.9 (11.57) | 9.6 (38.25) | -3.5 (11.35) | -0.1 (42.41)
  QTcF; Day 71; n=2,13,5,21: number analyzed (Participants) | 2 | 13 | 5 | 21
  QTcF; Day 71; n=2,13,5,21 | -11.1 (27.30) | 7.6 (30.12) | -3.5 (18.48) | -1.2 (17.15)
  QTcF; Day 85; n=2,13,5,20: number analyzed (Participants) | 2 | 13 | 5 | 20
  QTcF; Day 85; n=2,13,5,20 | 2.5 (17.46) | 10.6 (28.46) | -7.0 (11.36) | 0.6 (12.45)

8. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Indicated Time Points
Description: SBP and DBP were measured in a supine or semi-supine position after approximately 5 minutes rest. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline (Day 1 pre-dose), Days 8, 15, 29, 43, 57, 71 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 15 | 5 | 25
Millimeters of Mercury (mmHg)
  SBP; Day 8; n=3,15,5,25 | -9.7 (5.69) | 0.5 (12.61) | -4.6 (14.33) | 2.7 (11.0)
  SBP; Day 15; n=3,15,5,25 | -2.0 (7.55) | -2.7 (11.21) | -13.0 (12.79) | 4.6 (9.43)
  SBP; Day 29; n=3,15,5,24: number analyzed (Participants) | 3 | 15 | 5 | 24
  SBP; Day 29; n=3,15,5,24 | -9.3 (15.70) | -0.8 (10.82) | -8.2 (19.12) | 1.9 (11.94)
  SBP; Day 43; n=3,14,5,24: number analyzed (Participants) | 3 | 14 | 5 | 24
  SBP; Day 43; n=3,14,5,24 | -7.0 (9.54) | -2.0 (15.11) | -11.4 (19.72) | -1.6 (10.01)
  SBP; Day 57; n=3,14,5,23: number analyzed (Participants) | 3 | 14 | 5 | 23
  SBP; Day 57; n=3,14,5,23 | -14.7 (17.21) | 0.5 (16.19) | -9.6 (18.49) | -0.3 (12.84)
  SBP; Day 71; n=3,14,5,23: number analyzed (Participants) | 3 | 14 | 5 | 23
  SBP; Day 71; n=3,14,5,23 | -7.0 (9.85) | 1.1 (14.35) | -8.2 (12.19) | 1.2 (14.40)
  SBP; Day 85; n=3,14,5,22: number analyzed (Participants) | 3 | 14 | 5 | 22
  SBP; Day 85; n=3,14,5,22 | -4.3 (12.70) | -0.1 (14.68) | -4.8 (11.23) | 1.9 (12.97)
  DBP; Day 8; n=3,15,5,25 | 2.00 (5.00) | 2.0 (11.32) | 1.0 (8.69) | -0.4 (7.12)
  DBP; Day 15; n=3,15,5,25 | 0.3 (6.11) | 0.3 (7.85) | 0.4 (4.39) | 1.1 (7.61)
  DBP; Day 29; n=3,15,5,24: number analyzed (Participants) | 3 | 15 | 5 | 24
  DBP; Day 29; n=3,15,5,24 | -4.0 (8.89) | 0.2 (8.28) | -2.0 (6.04) | 0.7 (7.65)
  DBP; Day 43; n=3,14,5,24: number analyzed (Participants) | 3 | 14 | 5 | 24
  DBP; Day 43; n=3,14,5,24 | 0.3 (14.36) | -0.3 (8.96) | -1.4 (8.76) | -0.8 (6.68)
  DBP; Day 57; n=3,14,5,23: number analyzed (Participants) | 3 | 14 | 5 | 23
  DBP; Day 57; n=3,14,5,23 | -3.7 (8.33) | 0.8 (9.90) | 1.4 (6.43) | -0.9 (7.78)
  DBP; Day 71; n=3,14,5,23: number analyzed (Participants) | 3 | 14 | 5 | 23
  DBP; Day 71; n=3,14,5,23 | -7.0 (9.17) | 1.4 (8.36) | -7.2 (9.76) | -1.5 (6.90)
  DBP; Day 85; n=3,14,5,22: number analyzed (Participants) | 3 | 14 | 5 | 22
  DBP; Day 85; n=3,14,5,22 | 1.0 (6.24) | 2.1 (10.79) | -1.4 (7.67) | -0.4 (7.50)

9. Primary Outcome: Change From Baseline in Respiratory Rate at Indicated Time Points
Description: Respiratory rate was measured in a supine or semi-supine position after approximately 5 minutes rest. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline (Day 1 pre-dose), Days 8, 15, 29, 43, 57, 71 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 15 | 5 | 25
Breaths per minute
  Day 8; n=3,15,5,25 | 0.7 (1.53) | 0.1 (1.13) | -0.4 (2.61) | 0.0 (1.14)
  Day 15; n=3,15,5,25 | 1.0 (1.73) | 0.2 (1.08) | -1.2 (1.79) | 0.2 (1.91)
  Day 29; n=3,15,5,24: number analyzed (Participants) | 3 | 15 | 5 | 24
  Day 29; n=3,15,5,24 | 1.0 (1.00) | -0.2 (1.47) | -1.6 (1.67) | 0.1 (1.28)
  Day 43; n=3,14,5,24: number analyzed (Participants) | 3 | 14 | 5 | 24
  Day 43; n=3,14,5,24 | 1.7 (0.58) | 0.3 (1.33) | -0.8 (1.10) | 0.5 (2.70)
  Day 57; n=3,14,5,23: number analyzed (Participants) | 3 | 14 | 5 | 23
  Day 57; n=3,14,5,23 | 1.7 (2.08) | 0.2 (0.70) | 0.4 (3.29) | 0.6 (2.00)
  Day 71; n=3,14,5,23: number analyzed (Participants) | 3 | 14 | 5 | 23
  Day 71; n=3,14,5,23 | 1.7 (0.58) | 0.5 (0.65) | 0.0 (2.45) | 0.7 (2.07)
  Day 85; n=3,14,5,22: number analyzed (Participants) | 3 | 14 | 5 | 22
  Day 85; n=3,14,5,22 | 0.7 (0.58) | 0.4 (0.84) | -0.4 (2.61) | 0.5 (1.60)

10. Primary Outcome: Change From Baseline in Body Temperature at Indicated Time Points
Description: Body temperature was measured in a supine or semi-supine position after approximately 5 minutes rest. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline (Day 1 pre-dose), Days 8, 15, 29, 43, 57, 71 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 15 | 5 | 25
Degrees Celsius
  Day 8; n=3,15,5,25 | 0.60 (0.529) | -0.03 (0.209) | -0.06 (0.261) | 0.06 (0.222)
  Day 15; n=3,15,5,25 | 0.80 (0.500) | -0.07 (0.171) | -0.04 (0.219) | 0.06 (0.251)
  Day 29; n=3,15,5,24: number analyzed (Participants) | 3 | 15 | 5 | 24
  Day 29; n=3,15,5,24 | 0.60 (0.656) | -0.02 (0.204) | 0.10 (0.187) | 0.11 (0.249)
  Day 43; n=3,14,5,24: number analyzed (Participants) | 3 | 14 | 5 | 24
  Day 43; n=3,14,5,24 | 0.53 (0.513) | -0.01 (0.251) | 0.04 (0.270) | 0.06 (0.286)
  Day 57; n=3,14,5,23: number analyzed (Participants) | 3 | 14 | 5 | 23
  Day 57; n=3,14,5,23 | 0.53 (0.462) | -0.02 (0.226) | -0.02 (0.239) | 0.16 (0.310)
  Day 71; n=3,14,5,23: number analyzed (Participants) | 3 | 14 | 5 | 23
  Day 71; n=3,14,5,23 | 0.27 (0.404) | -0.06 (0.210) | -0.00 (0.141) | 0.17 (0.255)
  Day 85; n=3,14,5,22: number analyzed (Participants) | 3 | 14 | 5 | 22
  Day 85; n=3,14,5,22 | 0.53 (0.379) | -0.10 (0.162) | -0.12 (0.356) | 0.14 (0.353)

11. Primary Outcome: Change From Baseline in Vital Sign-heart Rate at Indicated Time Points
Description: Vital sign-heart rate was planned to be assessed as a measure of safety and tolerability.
Time Frame: Baseline (Day 1 pre-dose), Days 8, 15, 29, 43, 57, 71 and 85
Population: The data for assessment of vital sign-heart rate was not collected.
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Pre-dose Plasma Concentrations of GSK2982772 on Days 8 and 43
Description: Blood samples were collected on Day 8 and Day 43 for determining pre-dose plasma concentrations of GSK2982772. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: Pre-dose on Day 8 and Day 43
Population: Pharmacokinetic GSK298772 Population comprised of participants in the safety population who received an active dose and for whom a GSK2982772 pharmacokinetic sample was obtained and analyzed. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 5 | 24
Nanogram per milliliter
  Day 8;n=5,24 | 88.332 (96.5705) | 181.774 (322.8428)
  Day 43;n=5,23: number analyzed (Participants) | 5 | 23
  Day 43;n=5,23 | 33.994 (51.1033) | 142.792 (176.2630)

13. Secondary Outcome: Post-dose Plasma Concentrations of GSK2982772 on Days 1, 8, and 43 at 1, 2, 4 and 6 Hours
Description: Blood samples were collected on Day 1, Day 8 and Day 43 for determining post-dose plasma concentrations of GSK2982772. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: Days 1, 8 and 43: 1, 2, 4 and 6 hours post-dose
Population: Pharmacokinetic GSK298772 Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 5 | 27
Nanogram per milliliter
  Day 1;1 hour;n=5,27 | 851.000 (375.5110) | 953.037 (556.4630)
  Day 1;2 hour;n=5,27 | 656.000 (386.5741) | 911.630 (376.7128)
  Day 1;4 hour;n=5,27 | 269.600 (156.3052) | 421.215 (211.7969)
  Day 1;6 hour;n=5,27 | 120.240 (54.6881) | 382.419 (485.6076)
  Day 8;1 hour;n=5,23: number analyzed (Participants) | 5 | 23
  Day 8;1 hour;n=5,23 | 796.600 (397.7120) | 881.783 (550.4666)
  Day 8;2 hour;n=5,24: number analyzed (Participants) | 5 | 24
  Day 8;2 hour;n=5,24 | 689.000 (317.5602) | 930.958 (446.0379)
  Day 8;4 hour;n=5,24: number analyzed (Participants) | 5 | 24
  Day 8;4 hour;n=5,24 | 265.000 (129.6360) | 520.958 (324.4127)
  Day 8;6 hour;n=5,23: number analyzed (Participants) | 5 | 23
  Day 8;6 hour;n=5,23 | 112.280 (78.0491) | 444.470 (358.1685)
  Day 43;1 hour;n=5,23: number analyzed (Participants) | 5 | 23
  Day 43;1 hour;n=5,23 | 672.200 (165.4470) | 862.487 (501.4882)
  Day 43;2 hour;n=5,23: number analyzed (Participants) | 5 | 23
  Day 43;2 hour;n=5,23 | 598.600 (253.0036) | 872.652 (354.1155)
  Day 43;4 hour;n=5,23: number analyzed (Participants) | 5 | 23
  Day 43;4 hour;n=5,23 | 313.200 (226.0845) | 553.783 (430.5811)
  Day 43;6 hour;n=5,23: number analyzed (Participants) | 5 | 23
  Day 43;6 hour;n=5,23 | 177.980 (192.6731) | 332.522 (240.9716)

14. Secondary Outcome: Trough Plasma Concentration of GSK2982772 on Day 85
Description: Blood samples were collected to evaluate plasma concentration of GSK2982772. Pharmacokinetic parameters including trough plasma concentration was determined using standard non-compartmental methods.
Time Frame: Day 85
Population: Pharmacokinetic GSK298772 Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 5 | 17
Nanogram per milliliter | 54.64 (50.714) | 391.11 (694.270)

15. Secondary Outcome: Pre-dose Plasma Concentrations of Methotrexate on Days 1, 8 and 43
Description: Blood samples were collected on Day 1, Day 8 and Day 43 for determining pre-dose plasma concentrations of methotrexate. Pharmacokinetic parameters were determined using standard non-compartmental methods. Only participants who received methotrexate during the study were included.
Time Frame: Pre-dose on Days 1, 8 and 43
Population: Pharmacokinetic Methotrexate Population comprised of participants in the safety population who received an active dose and for whom a methotrexate pharmacokinetic sample was obtained and analyzed. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 13 | 5 | 22
Nanogram per milliliter
  Day 1;n=3,13,5,22 | 0.450 (0.7794) | 16.236 (56.4280) | 0.546 (0.7909) | 6.309 (15.4993)
  Day 8;n=3,12,5,17: number analyzed (Participants) | 3 | 12 | 5 | 17
  Day 8;n=3,12,5,17 | 1.117 (1.9341) | 0.509 (0.9879) | 4.640 (10.3754) | 11.939 (47.4493)
  Day 43;n=3,11,5,19: number analyzed (Participants) | 3 | 11 | 5 | 19
  Day 43;n=3,11,5,19 | 36.000 (62.3538) | 0.909 (2.0658) | 1.512 (3.3809) | 1.445 (3.1606)

16. Secondary Outcome: Percent Change From Baseline in C-Reactive Protein (CRP)
Description: CRP is an inflammatory biomarker present in blood. Blood samples were collected at indicated time points for the assessment of CRP. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Percent change from Baseline was calculated by 100*[(post-dose value minus Baseline value)/ Baseline value].
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 14 | 5 | 24
Percent change
  Day 43;n=3,14,5,24 | -24.02 (53.259) | 63.02 (331.286) | -10.37 (94.318) | 12.68 (107.207)
  Day 85;n=3,14,5,22: number analyzed (Participants) | 3 | 14 | 5 | 22
  Day 85;n=3,14,5,22 | -43.62 (49.968) | 220.05 (828.334) | -16.42 (70.096) | 274.25 (879.900)

17. Secondary Outcome: Percent Change From Baseline in Interleukin 6 (IL6)
Description: IL6 is an inflammatory biomarker present in blood. Blood samples were collected at indicated time points for the assessment of IL6. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Percent change from Baseline was calculated by 100*[(post-dose value minus Baseline value)/ Baseline value].
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 14 | 5 | 24
Percent change
  Day 43;n=3,14,5,24 | 89.12 (96.649) | 55.00 (257.661) | -3.95 (66.008) | 74.49 (358.187)
  Day 85;n=3,14,5,22: number analyzed (Participants) | 3 | 14 | 5 | 22
  Day 85;n=3,14,5,22 | 5.21 (16.978) | 27.52 (97.215) | -24.44 (67.817) | 0.52 (106.029)

18. Secondary Outcome: Percent Change From Baseline in Matrix Metalloproteinase-1 (MMP-1), MMP-3, and MMP-13
Description: MMP-1, MMP-3, and MMP-13 are an inflammatory biomarkers present in blood. Blood samples were collected at indicated time points for the assessment of MMP-1, MMP-3, and MMP-13. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Percent change from Baseline was calculated by 100*[(post-dose value minus Baseline value)/ Baseline value].
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 14 | 5 | 24
Percent change
  MMP-1;Day 43;n=3,14,5,24 | -11.25 (6.591) | -4.04 (23.016) | -15.36 (13.399) | -4.07 (27.244)
  MMP-1;Day 85;n=3,14,5,22: number analyzed (Participants) | 3 | 14 | 5 | 22
  MMP-1;Day 85;n=3,14,5,22 | -19.77 (28.013) | 9.75 (41.645) | -20.21 (19.417) | -1.61 (28.420)
  MMP-3;Day 43;n=3,14,5,24 | 8.86 (27.501) | 6.07 (27.883) | -26.82 (20.757) | -4.07 (36.176)
  MMP-3;Day 85;n=3,14,5,22: number analyzed (Participants) | 3 | 14 | 5 | 22
  MMP-3;Day 85;n=3,14,5,22 | 32.61 (32.849) | 11.98 (42.337) | -38.26 (19.306) | -2.14 (34.751)
  MMP-13;Day 43;n=3,12,5,22: number analyzed (Participants) | 3 | 12 | 5 | 22
  MMP-13;Day 43;n=3,12,5,22 | -6.45 (7.000) | 32.94 (139.157) | -7.27 (34.373) | -3.55 (29.506)
  MMP-13;Day 85;n=3,11,5,17: number analyzed (Participants) | 3 | 11 | 5 | 17
  MMP-13;Day 85;n=3,11,5,17 | -34.65 (35.926) | 114.18 (223.386) | -21.16 (31.372) | 67.91 (157.027)

19. Secondary Outcome: Percent Change From Baseline in Tissue Inhibitor of Metalloproteinases-1 (TIMP-1)
Description: TIMP-1 is an inflammatory biomarker present in blood. Blood samples were collected at indicated time points for the assessment of TIMP-1. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Percent change from Baseline was calculated by 100*[(post-dose value minus Baseline value)/ Baseline value].
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 14 | 5 | 24
Percent change
  Day 43;n=3,14,5,24 | -1.82 (6.578) | -9.89 (37.032) | -7.39 (11.298) | -5.59 (23.922)
  Day 85;n=3,14,5,22: number analyzed (Participants) | 3 | 14 | 5 | 22
  Day 85;n=3,14,5,22 | 35.61 (73.383) | -2.63 (57.144) | 49.38 (114.161) | -1.75 (33.789)

20. Secondary Outcome: Percent Change From Baseline in Monocyte Chemo Attractant Protein-1 (MCP-1)
Description: MCP-1 is an inflammatory biomarker present in blood. Blood samples were collected at indicated time points for the assessment of MCP-1. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Percent change from Baseline was calculated by 100*[(post-dose value minus Baseline value)/ Baseline value].
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 14 | 5 | 23
Percent change
  Day 43;n=3,14,5,23 | -4.57 (19.262) | 388.23 (565.617) | -4.37 (11.309) | 156.79 (297.549)
  Day 85;n=3,14,5,21: number analyzed (Participants) | 3 | 14 | 5 | 21
  Day 85;n=3,14,5,21 | -33.39 (49.411) | 422.45 (514.842) | -30.35 (36.118) | 199.94 (392.590)

21. Secondary Outcome: Percent Change From Baseline in Migration Inhibitory Factor (MIF)
Description: MIF is an inflammatory biomarker present in blood. Blood samples were collected at indicated time points for the assessment of MIF. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Percent change from Baseline was calculated by 100*[(post-dose value minus Baseline value)/ Baseline value].
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 14 | 5 | 24
Percent change
  Day 43;n=3,14,5,24 | 8.98 (29.041) | 4.69 (46.772) | 120.23 (362.931) | 34.46 (160.400)
  Day 85;n=3,14,5,22: number analyzed (Participants) | 3 | 14 | 5 | 22
  Day 85;n=3,14,5,22 | 15.39 (26.888) | -15.72 (49.080) | -11.80 (47.351) | -5.76 (49.377)

22. Secondary Outcome: Percent Change From Baseline in Myeloid-related Protein 8/14 (MRP8/14)
Description: MRP8/14 is an inflammatory biomarker present in blood. Blood samples were collected at indicated time points for the assessment of MRP8/14. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Percent change from Baseline was calculated by 100*[(post-dose value minus Baseline value)/ Baseline value].
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 14 | 5 | 24
Percent change
  Day 43;n=3,14,5,24 | 3.15 (47.472) | 25.14 (75.189) | -49.21 (19.168) | -22.95 (38.992)
  Day 85;n=3,14,5,22: number analyzed (Participants) | 3 | 14 | 5 | 22
  Day 85;n=3,14,5,22 | 13.84 (66.492) | 70.37 (199.467) | -28.27 (17.112) | -11.35 (77.927)

23. Secondary Outcome: Change From Baseline in Bone Erosion Total Score by "Outcome Measures in Rheumatology, Rheumatoid Arthritis Magnetic Resonance Image Scoring System (OMERACT-RAMRIS)" Scoring System
Description: A total of 25 locations in the hand and wrist were evaluated for RAMRIS bone erosions. Individual location scores range from 0 (no erosions) to 10 (91 to 100 percent of bone eroded) based on the proportion of eroded bone compared to the "assessed bone volume" on all available images. The final bone erosion score was the sum of the individual location scores. The total score from the 25 locations ranges from 0 to 250, with 0 implying no bone erosion and 250 implying 91 to 100 percent bone eroded. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 13 | 5 | 24
Scores on a scale
  Day 43;n=3,13,5,24 | 0.7 (1.15) | 0.6 (1.04) | 0.4 (1.52) | -0.2 (1.83)
  Day 85;n=3,13,5,22: number analyzed (Participants) | 3 | 13 | 5 | 22
  Day 85;n=3,13,5,22 | 1.7 (2.89) | 1.3 (2.43) | 0.4 (1.52) | -0.1 (2.21)

24. Secondary Outcome: Change From Baseline in Bone Erosions by the Rheumatoid Arthritis MRI Quantitative (RAMRIQ) Scoring System
Description: RAMRIQ bone erosions (normalized) was a quantitative measurement from the bones and synovial capsules of the joints from the most affected (or dominant hand if equally affected). It was calculated as the sum of the individual measurements of the volume of bone erosions divided by sum of the individual measurements of the bone volume. The total score ranged from 0 to 1, with 0 implying no erosive damage. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 13 | 5 | 23
Scores on a scale
  Day 43;n=2,13,5,23: number analyzed (Participants) | 2 | 13 | 5 | 23
  Day 43;n=2,13,5,23 | -0.00160 (0.002550) | -0.00110 (0.002265) | -0.00072 (0.001662) | -0.00069 (0.004145)
  Day 85;n=2,13,5,21: number analyzed (Participants) | 2 | 13 | 5 | 21
  Day 85;n=2,13,5,21 | -0.00069 (0.001134) | -0.00075 (0.001301) | -0.00273 (0.003505) | 0.00059 (0.003946)

25. Secondary Outcome: Change From Baseline in Bone Erosions by Modified Cartilage Loss Scoring System (CARLOS)
Description: Change from Baseline in bone erosions was planned to be assessed by modified CARLOS.
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: Safety Population. Data was not collected for this outcome measure, as bone erosion is not a part of modified CARLOS. Bone erosion was measured by OMERACT-RAMRIS and RAMRIQ scoring system and is presented in outcome measures 23 and 24, respectively.
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 0 | 0 | 0 | 0

26. Secondary Outcome: Change From Baseline in Synovitis by OMERACT-RAMRIS Scoring System
Description: A total of 8 joints in the hand and wrist were evaluated for RAMRIS synovitis. Individual joint scores were assessed on a scale of 0 (no synovitis) to 3 (67 to 100 percent volume enhancement). The final synovitis score was the sum of the individual joint scores. The total score from 8 joints ranges from 0 to 24, with 0 implying normal (no synovitis) and 24 implying 67 to 100 percent volume enhancement. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 13 | 5 | 24
Scores on a scale
  Day 43;n=3,13,5,24 | 0.0 (1.73) | 0.3 (1.55) | -0.4 (1.52) | -0.3 (1.90)
  Day 85;n=3,13,5,22: number analyzed (Participants) | 3 | 13 | 5 | 22
  Day 85;n=3,13,5,22 | 0.3 (1.15) | 0.5 (2.67) | -0.4 (1.52) | -0.5 (2.20)

27. Secondary Outcome: Change From Baseline in Synovitis by RAMRIQ Scoring System
Description: RAMRIQ synovitis (normalised) was a quantitative measurement from the bones and synovial capsules of the joints from the most affected (or dominant hand if equally affected). It was calculated as the sum of the individual measurements of the volume of enhancing pannus (VEP) divided by sum of the individual measurements of the joint volume. The total score ranged from 0 to 1, with 0 implying no synovitis. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 2 | 13 | 5 | 23
Scores on a scale
  Day 43;n=2,13,5,23 | -0.0570 (0.02302) | -0.0165 (0.04302) | -0.0592 (0.06931) | -0.0084 (0.10490)
  Day 85;n=2,13,5,21: number analyzed (Participants) | 2 | 13 | 5 | 21
  Day 85;n=2,13,5,21 | -0.0659 (0.01625) | 0.0251 (0.12286) | -0.0270 (0.07061) | -0.0107 (0.11472)

28. Secondary Outcome: Change From Baseline in Synovitis by Modified CARLOS
Description: Change from Baseline in synovitis was planned to be assessed by modified CARLOS.
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: Safety Population. Data was not collected for this outcome measure, as synovitis is not a part of modified CARLOS. Synovitis was measured by OMERACT-RAMRIS and RAMRIQ scoring system and is presented in outcome measures 26 and 27, respectively.
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 0 | 0 | 0 | 0

29. Secondary Outcome: Change From Baseline in Bone Edema by OMERACT-RAMRIS Scoring System
Description: A total of 25 locations in the hand and wrist were evaluated for RAMRIS bone edema or osteitis. Individual location scores range from 0 (no edema) to 3 (67 to 100 percent involvement of original articular bone) based on the proportion of estimated originally non-eroded bone involved. The final bone edema or osteitis score is the sum of the individual location scores. The total score from the 25 locations ranges from 0 to 75, with 0 implying no bone edema or osteitis and 75 implying 67 to 100 percent involvement of original articular bone. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 13 | 5 | 24
Scores on a scale
  Day 43;n=3,13,5,24 | -1.0 (1.73) | -0.2 (1.52) | -0.8 (3.27) | -0.9 (2.47)
  Day 85;n=3,13,5,22: number analyzed (Participants) | 3 | 13 | 5 | 22
  Day 85;n=3,13,5,22 | 0.3 (0.58) | 0.3 (1.38) | -4.4 (6.80) | -1.1 (2.59)

30. Secondary Outcome: Change From Baseline in Bone Edema by RAMRIQ Scoring System
Description: RAMRIQ bone edema (normalised) was a quantitative measurement from the bones and synovial capsules of the joints from the most affected (or dominant hand if equally affected). It was calculated as the sum of the individual measurements of the Volume of bone edema divided by sum of the individual measurements of the bone volume. The total score ranged from 0 to 1, with 0 implying no bone marrow lesions. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 2 | 13 | 5 | 22
Scores on a scale
  Day 43;n=2,13,5,22 | -0.00396 (0.000647) | -0.00463 (0.007465) | -0.01963 (0.031481) | -0.00095 (0.018745)
  Day 85;n=2,13,5,21: number analyzed (Participants) | 2 | 13 | 5 | 21
  Day 85;n=2,13,5,21 | 0.00116 (0.010166) | -0.00229 (0.010143) | -0.03921 (0.055431) | -0.00384 (0.016126)

31. Secondary Outcome: Change From Baseline in Bone Edema by Modified CARLOS
Description: Change from Baseline in bone edema was planned to be assessed by modified CARLOS.
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: Safety Population. Data was not collected for this outcome measure, as bone edema is not a part of modified CARLOS. Bone edema was measured by OMERACT-RAMRIS and RAMRIQ scoring system and is presented in outcome measures 29 and 30, respectively.
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 0 | 0 | 0 | 0

32. Secondary Outcome: Change From Baseline in Joint Space Narrowing by OMERACT-RAMRIS Scoring System
Description: Change from Baseline in joint space narrowing was planned to be assessed by OMERACT-RAMRIS scoring system.
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: Safety Population. Data was not collected for this outcome measure, as joint space narrowing is not a part of OMERACT-RAMRIS scoring system. Joint space narrowing was measured by RAMRIQ scoring system and modified CARLOS and is presented in outcome measures 33 and 34, respectively.
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 0 | 0 | 0 | 0

33. Secondary Outcome: Change From Baseline in Joint Space Narrowing by RAMRIQ Scoring System
Description: RAMRIQ joint space narrowing was a quantitative measurement from the bones and synovial capsules of the joints from the most affected (or dominant hand if equally affected). It was calculated as the sum of the individual measurements (in millimeter) for the joints measured. The minimum possible total score is 0 implying complete loss of the joint space. The maximum possible total score will be largest possible joint space. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 2 | 13 | 5 | 23
Scores on a scale
  Day 43;n=2,13,5,23 | 1.121 (1.4793) | 0.378 (1.3394) | 0.484 (2.8980) | -0.335 (1.4365)
  Day 85;n=2,13,5,21: number analyzed (Participants) | 2 | 13 | 5 | 21
  Day 85;n=2,13,5,21 | 0.534 (0.8910) | 0.216 (0.6974) | 0.235 (2.2525) | -0.433 (1.1205)

34. Secondary Outcome: Change From Baseline in Joint Space Narrowing by Modified CARLOS
Description: A total of 20 locations in the hand and wrist were evaluated for CARLOS joint space narrowing/cartilage loss. Individual location scores range from 0 (no cartilage loss or Joint Space Narrowing) to 4 (complete ankylosis) in increments of 0.5 based on the amount of narrowing present in a given joint. The final cartilage loss score was the sum of the individual location scores. The total score from 20 location ranged from 0 to 80, with 0 implying no cartilage loss at any location and 80 implying complete ankylosis. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 13 | 5 | 24
Scores on a scale
  Day 43;n=3,13,5,24 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.08 (0.408)
  Day 85;n=3,13,5,22: number analyzed (Participants) | 3 | 13 | 5 | 22
  Day 85;n=3,13,5,22 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.09 (0.426)

35. Secondary Outcome: Change From Baseline in Exchange Rate (Ktrans)
Description: Contrast agent volume transfer constant (Ktrans) relates to the exchange of contrast agent between the blood plasma and the tissue extravascular extracellular spaces and reflects blood flow and capillary permeability. Ktrans was measured by dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) tracer kinetic modeling in the most affected hand/wrist at indicated time points. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Per minute
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 2 | 9 | 5 | 19
Per minute
  Day 43;n=2,9,5,19 | 0.0012 (0.00076) | 0.0022 (0.01214) | -0.0095 (0.01716) | -0.0018 (0.01443)
  Day 85;n=2,9,5,17: number analyzed (Participants) | 2 | 9 | 5 | 17
  Day 85;n=2,9,5,17 | 0.0002 (0.01726) | -0.0021 (0.01385) | -0.0073 (0.00618) | -0.0043 (0.01747)

36. Secondary Outcome: Change From Baseline in Interstitial Volume (Ve)
Description: Interstitial volume (Ve) is the fractional volume of the extravascular extracellular (EC) space per unit volume tissue within which contrast agent can accumulate. Ve was measured by DCE-MRI in most affected hand/wrist at indicated time points. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio of EC space to tissue volume
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 2 | 9 | 5 | 18
Ratio of EC space to tissue volume
  Day 43;n=2,9,5,18 | -0.305 (0.3128) | -0.066 (0.3615) | -0.140 (0.4825) | 0.073 (0.4044)
  Day 85;n=2,9,5,15: number analyzed (Participants) | 2 | 9 | 5 | 15
  Day 85;n=2,9,5,15 | 0.009 (0.7840) | -0.024 (0.2450) | -0.278 (0.5170) | 0.113 (0.4664)

37. Secondary Outcome: Change From Baseline in Fractional Volume of Blood Plasma (Vp)
Description: Fractional volume of blood plasma (Vp) is the fractional volume of blood plasma per unit volume of tissue. Vp was measured by DCE-MRI in most affected hand/wrist at indicated time points. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio of plasma volume to tissue volume
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 2 | 9 | 5 | 19
Ratio of plasma volume to tissue volume
  Day 43;n=2,9,5,19 | 0.0018 (0.00166) | 0.0007 (0.00678) | -0.0023 (0.00786) | -0.0007 (0.00358)
  Day 85;n=2,9,5,17: number analyzed (Participants) | 2 | 9 | 5 | 17
  Day 85;n=2,9,5,17 | 0.0000 (0.00019) | -0.0022 (0.00407) | -0.0001 (0.00272) | -0.0007 (0.00282)

38. Secondary Outcome: Change From Baseline in Initial Rate of Enhancement (IRE)
Description: Initial Rate of Enhancement (IRE) is a measure of how quickly tissue enhances over 60 seconds following administration of contrast agent. IRE was measured by DCE-MRI in most affected hand/wrist at indicated time points. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Millimole per second
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 2 | 9 | 5 | 19
Millimole per second
  Day 43;n=2,9,5,19 | -0.00002 (0.000044) | 0.00008 (0.000538) | -0.00043 (0.000750) | -0.00008 (0.000575)
  Day 85;n=2,9,5,17: number analyzed (Participants) | 2 | 9 | 5 | 17
  Day 85;n=2,9,5,17 | -0.00011 (0.000566) | -0.00010 (0.000542) | -0.00037 (0.000271) | -0.00014 (0.000735)

39. Secondary Outcome: Change From Baseline in Maximal Signal Intensity Enhancement (ME)
Description: Maximum enhancement (ME) is a measure of the maximum concentration of contrast agent in the tissue over the duration of the DCE-MRI time series. ME was measured by DCE-MRI in most affected hand/wrist at indicated time points. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Millimole
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 2 | 9 | 5 | 19
Millimole
  Day 43;n=2,9,5,19 | -0.0300 (0.00994) | 0.0029 (0.05405) | -0.0531 (0.06876) | 0.0007 (0.06159)
  Day 85;n=2,9,5,17: number analyzed (Participants) | 2 | 9 | 5 | 17
  Day 85;n=2,9,5,17 | -0.0533 (0.00473) | -0.0138 (0.05168) | -0.0584 (0.06009) | -0.0074 (0.07180)

40. Secondary Outcome: Change From Baseline in Disease Activity Score 28-C-Reactive Protein (DAS28-CRP) Scores
Description: The DAS28-CRP is a composite measure of inflammation in rheumatoid arthritis calculated from the sum of tender joint count 28 (TJC28), swollen joint count (SJC28), CRP and patient global assessment of disease activity (PtGA). The formula used to calculate DAS28 score was 0.56 multiplied by square root of TJC28 plus 0.28 multiplied by square root of SJC28 plus 0.36 log of (CRP plus 1) plus 0.014 multiplied by PtGA plus 0.96. Scores of DAS28-CRP ranged from 0.96 to 9.4 with higher scores indicating greater disease burden. A DAS28-CRP score of <=2.6 suggested remission, <3.2 suggested a low level of disease activity, while a score of >5.1 suggested a high level of disease activity. Baseline was defined as the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Day 85
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 12 | 5 | 22
Scores on a scale | -1.00 [-2.45 to 0.46] | -0.87 [-1.57 to -0.17] | -1.47 [-2.60 to 0.35] | -1.23 [-1.75 to 0.71]

41. Secondary Outcome: Number of Participants Achieving Categorical DAS28-CRP Response Using European League Against Rheumatism [EULAR] Response
Description: DAS28-CRP scores were categorized using EULAR response criteria. Response at a given time point was defined based on the combination of current DAS28 score and the improvement in the current DAS28 score relative to Baseline. The definition of no response, moderate response and good response was as; if current DAS28 <=3.2 and DAS28 decrease from Baseline (>1.2: good response), (>0.6 to <=1.2: moderate response) and (<=0.6: no response); if current DAS28 >3.2 to <=5.1 and DAS28 decrease from Baseline value (>1.2: moderate response), (>0.6 to <=1.2: moderate response) and (<=0.6: no response) and if current DAS28 >5.1 and DAS28 decrease from Baseline value (>1.2: moderate response), (>0.6 to <=1.2: no response) and (<=0.6: no response). If the post-Baseline DAS28-CRP score was missing, then the corresponding EULAR category was set to missing.
Time Frame: Day 85
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 12 | 5 | 22
Participants
  No response | 2 | 6 | 1 | 7
  Moderate response | 0 | 4 | 2 | 8
  Good response | 1 | 2 | 2 | 7

42. Secondary Outcome: Number of Participants Achieving Categorical American College of rheumatology20/50/70 (ACR20/50/70) Response
Description: The ACR score was based on improvement from Baseline in tender joint counts and swollen joint counts. A participant had achieved ACR20 if he experienced >=20 percent improvement from Baseline in Tender Joint count 28 (TJC28) and Swollen Joint Count 28 (SJC28) and a >=20 percent improvement from Baseline in 3 out of 5 of the following assessments: participant pain assessment on a 100 millimeter (mm) visual analog scale (VAS), participant global assessment on a 100 mm VAS scale, physician global assessment on a 100 mm VAS scale, C-reactive protein and Health Assessment Questionnaire - Disability Index (HAQ-DI). Similarly, ACR50 and ACR70 are calculated using 50 or 70 percent improvement from baseline respectively. For all visits, if any of the component scores were missing; then those scores were considered as not having met the criteria for improvement.
Time Frame: Day 85
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 3 | 15 | 5 | 28
Participants
  ACR20 | 1 | 6 | 3 | 12
  ACR50 | 1 | 2 | 0 | 5
  ACR70 | 1 | 1 | 0 | 4

43. Other Pre Specified Outcome: Change From Baseline in Joint Volume
Description: Joint volume was planned to be measured by DCE-MRI in most affected hand/wrist at indicated time points.
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: Safety Population. This was an other pre-specified outcome measure. Data will not be analyzed and reported.
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 0 | 0 | 0 | 0

44. Other Pre Specified Outcome: Change From Baseline in Enhancing Volume
Description: Enhancing volume was planned to be measured by DCE-MRI in most affected hand/wrist at indicated time points.
Time Frame: Baseline (Day 1 pre-dose), Days 43 and 85
Population: Safety Population. This was an other pre-specified outcome measure. Data will not be analyzed and reported.
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: On-therapy non-SAEs and SAEs were reported from start of study treatment and up to 112 days
Description: Non-SAE and SAEs were reported for Safety Population. Adverse events were presented treatment-wise.
Groups:
- GSK2982772 60mg BID: Participants received GSK2982772 orally twice daily (BID) for 84 days (12 weeks). Participants received methotrexate for the treatment of RA during conduct of the study, if required.
- GSK2982772 60mg TID: Participants received GSK2982772 orally three times daily (TID) (approximately 8 hours apart) for 84 days (12 weeks). Participants received methotrexate for the treatment of RA during conduct of the study, if required.
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60mg BID | GSK2982772 60mg TID
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/15 | 0/5 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/15 | 0/5 | 2/28
Other Adverse Events (participants affected / at risk) | 3/3 | 10/15 | 3/5 | 16/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo BID (N=3) | Placebo TID (N=15) | GSK2982772 60mg BID (N=5) | GSK2982772 60mg TID (N=28)
Retinal vein thrombosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo BID (N=3) | Placebo TID (N=15) | GSK2982772 60mg BID (N=5) | GSK2982772 60mg TID (N=28)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pertussis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-08-03): https://cdn.clinicaltrials.gov/large-docs/92/NCT02858492/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/92/NCT02858492/SAP_001.pdf